CLINICAL TRIAL: NCT01729455
Title: A 5-Year Prospective Observational Registry to Assess Adverse Events of Interest and Effectiveness in Adults With Active, Autoantibody-Positive Systemic Lupus Erythematosus Treated With or Without BENLYSTA™ (Belimumab)
Brief Title: Safety and Effectiveness of BENLYSTA (Belimumab) in Systemic Lupus Erythematosus (SLE) Registry
Acronym: SABLE
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116543; HGS1006-C1124 (Other: Human Genome Sciences Inc.)
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Belimumab; BENLYSTA; Systemic Lupus Erythematosus; Autoimmune Disease; Autoantibodies
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — belimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BENLYSTA cohort: Participants with active, autoantibody-positive SLE treated with BENLYSTA at Baseline.
  Interventions: Biological: BENLYSTA; Other: SLE treatment
- Comparison cohort: Participants with active, autoantibody-positive SLE treated without BENLYSTA at Baseline.
  Interventions: Other: SLE treatment

INTERVENTIONS:
Biological: BENLYSTA — As prescribed.
  Belimumab is a recombinant, human, IgG1λ monoclonal antibody for the treatment of systemic lupus erythematosus.
  Other Names: belimumab
  Groups: BENLYSTA cohort
Other: SLE treatment — As prescribed.
  At baseline, SLE treatment must include an immunosuppressant. During the registry, SLE treatment may include any of the following (alone or in combination): immunosuppressants, corticosteroids, antimalarials, other biologics, investigational agents for SLE, as clinically indicated.

SUMMARY:
The purpose of this prospective, observational cohort study is to evaluate the incidence of adverse events of special interest (AESI) and effectiveness in participants with active, autoantibody-positive SLE treated with and without BENLYSTA (belimumab). Participants will be enrolled into 1 of 2 cohorts: (1) BENLYSTA cohort: participants receiving or initiating BENLYSTA plus standard of care (SOC) at Baseline; (2) comparison cohort: participants not receiving BENLYSTA but receiving SOC at Baseline. After enrollment, changes in lupus medications, including starting or stopping BENLYSTA, are at the discretion of the physician, and all participants will continue to be followed regardless of changes in their lupus medicines until study completion. All participants will be assessed for AESI including serious infections, opportunistic infections and other infections of interest, malignancies, selected serious psychiatric events and mortality. Data will be collected at enrollment and at 6 month intervals for 5 years. BENLYSTA is a registered trademark of GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18 years or older.
* Have a clinical diagnosis of active SLE.
* Current or history of autoantibody-positive SLE.
* Must be treated with SLE therapy including BENLYSTA and/or immunosuppressants (for example, azathioprine, methotrexate, cyclophosphamide, mycophenolate, and biologics).
* Have the ability to understand the requirements of the study, provide written informed consent, including consent for the use and disclosure of research-related health information, and comply with the study data collection procedures.

Exclusion Criteria:

* Treatment with an investigational drug within one year of enrollment. Investigational drug applies to any drug not approved for sale in the country it is being used.
* Currently enrolled in a placebo-controlled BENLYSTA (belimumab) clinical trial or a continuation protocol where belimumab is used as an investigational agent.
* Participants who have a history of BENLYSTA exposure, but are not currently receiving BENLYSTA.
* Participants only receiving an anti-malarial for SLE.
* Participants only receiving steroids for SLE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with active autoantibody-positive SLE.
Sampling Method: Non-Probability Sample
Enrollment: 3138 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with AESI | Up to 5 years
  AESI including malignancies (excluding non-melanoma skin cancers), non-melanoma skin cancers (NMSC), mortality, serious infections, opportunistic infections and other infections of interest, and selected serious psychiatric events will be summarized.

OTHER OUTCOMES:
Number of participants with organ damage | Up to 5 years
  Organ damage will be assessed by System Lupus International Collaborating Clinics/American College of Rheumatology (SLICC/ACR) Damage Index (SDI). It is designed to capture items of irreversible organ damage present for at least 6 months occurring in participants with SLE regardless of exact cause. It consists of 12 organ system scales each having subscales which comprises of up to 6 components.
Number of participants with use of concomitant SLE medications | Up to 5 years
  Concomitant SLE medications including steroids are the medications used to treat SLE (immunosuppressants, anti-malarials, corticosteroids, biologics, and investigational agents for SLE).
Number of participants with hospitalizations | Up to 5 years
  An inpatient hospitalization is defined as an admission for greater than 24 hours. An admission for administration of medication or for routine or planned clinical procedures will not be considered a hospitalization. Dates of hospital admission and discharge, and whether the hospitalization was SLE-related will be collected, as available.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (154):
- United States (88):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Goodyear, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Prescott, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Murrieta, California
  - GSK Investigational Site, Pomona, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, West Hills, California
  - GSK Investigational Site, Danbury, Connecticut
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Orangeburg, Connecticut
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Palm Harbor, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Morton Grove, Illinois
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Eagan, Minnesota
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Tupelo, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Teaneck, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Roslyn, New York
  - GSK Investigational Site, Smithtown, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, New Bern, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Rocky Mount, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Edmond, Oklahoma
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Oklahoma City6, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Hixson, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Allen, Texas
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Nassau Bay, Texas
  - GSK Investigational Site, Round Rock, Texas
  - GSK Investigational Site, San Marcos, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Glendale, Wisconsin
  - GSK Investigational Site, Manitowoc, Wisconsin
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad autOnoma de Bueno
  - GSK Investigational Site, Paraná
- Austria (4):
  - GSK Investigational Site, Graz
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- GSK Investigational Site, Leuven, Belgium
- Canada (5):
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- France (4):
  - GSK Investigational Site, Bondy
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Strasbourg
- Germany (15):
  - GSK Investigational Site, Bad Bramstedt
  - GSK Investigational Site, Bad Nauheim
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Düsseldorf
  - GSK Investigational Site, Elmshorn
  - GSK Investigational Site, Halle
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Heidelberg
  - GSK Investigational Site, Jena
  - GSK Investigational Site, Kiel
  - GSK Investigational Site, Leipzig
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Püttlingen
  - GSK Investigational Site, Stuttgart
- Israel (8):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Nahariya
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
- Italy (7):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Siena
  - GSK Investigational Site, Udine
- GSK Investigational Site, Lisbon, Portugal
- Slovakia (3):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Piešťany
- Spain (14):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, BaracaldoVizcaya
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Las Palmas
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Toledo
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, VigoPontevedra
  - GSK Investigational Site, Villajoyosa
- GSK Investigational Site, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No